CLINICAL TRIAL: NCT01016704
Title: Reinforcing Therapist Performance
Acronym: RTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Bryan R. Garner, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTP-1; 1R01AA017625-01 (NIH)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Incentive (Experimental)
  Interventions: Behavioral: Incentive

INTERVENTIONS:
Behavioral: Incentive — Participants assigned to the experimental condition are reinforced via monetary incentives for demonstrating superior delivery of an evidence treatment to clients
  Arms: Incentive

SUMMARY:
The specific aims of the proposed study are to evaluate the effectiveness and cost-effectiveness of providing monetary incentives to therapists as a method to improve implementation of evidence-based treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must work at one of the participating demonstration sites funded by the Center for Substance Abuse Treatment to deliver the Adolescent Community Reinforcement Approach and/or Assertive Continuing Care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Target A-CRA | 14 weeks post intake
  Based on a review of recordings of actual client sessions is an indicator of whether or not clients received 10 or more of 12 specified treatment procedures within no less than seven treatment sessions.
A-CRA Competence | Monthly
  Based on review of a randomly selected session recording is an indicator of whether or not participants delivered at least one treatment procedure at or above the level of competence required as part of the certification process.

SECONDARY OUTCOMES:
Percent of days abstinent | 6 months post-intake
  Based on client self report is the percentage of days during the past 90 days that clients reported not using any alcohol or other drugs.
Pay-for-performance Cost-Effectiveness | First six months of study
  The cost per unit of Target A-CRA, A-CRA Competene, and Percentage of Days Abstient in the experimental condition relative to the control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan R Garner, Ph.D., Principal Investigator — Chestnut Health Systems
Locations (1):
- Lighthouse Institute, Chestnut Health Systems, Normal, Illinois, United States

REFERENCES:
- [Result] Garner BR, Godley SH, Bair CM. The impact of pay-for-performance on therapists' intentions to deliver high-quality treatment. J Subst Abuse Treat. 2011 Jul;41(1):97-103. doi: 10.1016/j.jsat.2011.01.012. Epub 2011 Feb 11. PMID 21315539
- [Derived] Garner BR, Lwin AK, Strickler GK, Hunter BD, Shepard DS. Pay-for-performance as a cost-effective implementation strategy: results from a cluster randomized trial. Implement Sci. 2018 Jul 4;13(1):92. doi: 10.1186/s13012-018-0774-1. PMID 29973280
- [Derived] Garner BR, Godley SH, Dennis ML, Hunter BD, Bair CM, Godley MD. Using pay for performance to improve treatment implementation for adolescent substance use disorders: results from a cluster randomized trial. Arch Pediatr Adolesc Med. 2012 Oct;166(10):938-44. doi: 10.1001/archpediatrics.2012.802. PMID 22893231